CLINICAL TRIAL: NCT00000830
Title: Intracellular Pharmacokinetics of Zidovudine Triphosphate in Maternal and Infant Cord Blood Mononuclear Cells.
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: ACTG 296
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1998-03

CONDITIONS: HIV Infections; Pregnancy
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Natural History

SUMMARY:
To determine the levels of zidovudine triphosphate ( AZT-TP ) in maternal and fetal cord blood mononuclear cells. To determine the ratio of AZT-TP to endogenous nucleoside triphosphate levels in maternal and fetal cells. To determine the extent of drug transfer through the feto/placental unit.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24

CONTACTS AND LOCATIONS:
Overall Officials: Fridland A, Study Chair; Flynn P, Study Chair
Locations (6):
- United States (5):
  - Univ of Medicine & Dentistry of New Jersey / Univ Hosp, Newark, New Jersey
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Mount Sinai Med Ctr / Pediatrics, New York, New York
  - Regional Med Ctr at Memphis, Memphis, Tennessee
  - Saint Jude Children's Research Hosp of Memphis, Memphis, Tennessee
- San Juan City Hosp, San Juan, Puerto Rico

REFERENCES:
- [Background] Rodman JH, Flynn PM, Robbins BL, Blanchard S, Jimenez E, Rodriguez J, Fridland A. Zidovudine pharmacokinetics and intracellular pharmacology of zidovudine in HIV-infected women and newborn infants. Conf Retroviruses Opportunistic Infect. 1999 Jan 31-Feb 4;6th:146 (abstract no 419)